CLINICAL TRIAL: NCT02787577
Title: The SLuMBER Study: The Sleep Lengthening and Metabolic Health, Body Composition, Energy Balance and Cardiovascular Risk Study
Brief Title: The Sleep Lengthening and Metabolic Health, Body Composition, Energy Balance and Cardiovascular Risk Study
Acronym: SLuMBER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SLuMBER Study 2016
Record Dates: First submitted 2016-04-05; First posted 2016-06-01 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2016-06

CONDITIONS: Sleep
Keywords: Sleep Duration; Sleep Quality; Body Composition; Energy Intake; Energy Expenditure; Energy Balance; Cardiovascular Risk
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep Lengthening (Experimental): The intervention group will receive a personalised sleep consultation session to lengthen sleep by 1-1.5 hours per night by targeting sleep hygiene using behaviour change techniques for 4 weeks.
  Interventions: Behavioral: Sleep Lengthening
- Control (No Intervention): The control group will be asked to resume their normal lifestyle.

INTERVENTIONS:
Behavioral: Sleep Lengthening — Behaviour change techniques targeting sleep hygiene
  Arms: Sleep Lengthening

SUMMARY:
Short sleep duration has been associated with increased risk of weight gain and development of non-communicable diseases. Sleep deprivation studies have suggested the link between restricted sleep and risk of adiposity and cardiometabolic dysregulation may be causal. However, the severity and acuteness of sleep restriction schedules in laboratory-based studies could hinder the ecological validity of the findings. The pragmatic way forward is to assess how improved sleep in habitually short sleepers impacts the aforementioned outcomes. This study assesses the feasibility of lengthening sleep in short sleepers, as well as how improved sleep duration and/or quality impact metabolic health, body composition, energy balance and cardiovascular risk.

DETAILED DESCRIPTION:
Research Questions

* Is it feasible to improve sleep duration and quality in habitually short sleepers under free-living conditions?
* What are the effects of improved sleep duration and quality on body composition, energy balance, dietary intake, and cardio-metabolic risk factors?

Hypothesis

- Improved sleep duration and/or quality in habitually short sleepers will result in improved energy balance, diet quality, body composition, and cardio-metabolic risk profile.

Aims

* To assess the feasibility of improving sleep duration and/or quality in habitually short sleepers using behavioural approaches and public health messages targeting sleep hygiene.
* To identify how improved sleep duration and/or quality affect energy balance, diet quality, body composition, and cardio-metabolic risk profile.

Objectives

1. To develop a sleep extension strategy using behaviour change techniques (BCTs) targeting sleep hygiene.
2. To recruit healthy adults who are habitually short sleepers and randomise eligible participants to an intervention and control group.
3. To assess the feasibility and effectiveness of the intervention.
4. To measure energy balance, diet quality, body composition and cardio-metabolic risk factors pre- and post-treatment in the intervention and control groups.
5. To assess whether the intervention had an effect on the aforementioned parameters by comparing the intervention endpoints to control as well as baseline measures.
6. To run the statistical analysis both on an intention-to-treat basis as well as per-protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults (18-64 years)
* Habitually short sleepers (5-<7 hours of sleep per night on average on weekdays) - this is self-reported at screening, and confirmed by actigraphy when baseline measurement is taken.
* BMI: 18.5 - <30

Exclusion Criteria:

* Diagnosed medical conditions such as:
* Cardiovascular disease
* Type 1 or Type 2 Diabetes Mellitus
* Cancer (excluding basal carcinoma) in the past five years
* Chronic renal or liver disease
* Inflammatory bowel disease
* Hypo/hyperthyroidism
* Sleep conditions:
* Chronic use of sleeping aid medication
* Insomnia (Insomnia Severity Index - ISI Questionnaire)
* Sleep apnoea (Berlin Questionnaire)
* Extreme Chronotype (HorneOstberg questionnaire)
* Pregnancy or lactation
* Weight change of >3 kg in the previous two months
* Previous or current high alcohol intake (>28 units/week for males and >21 units/week for females) or substance abuse
* Smoking
* Working hours outside 7 am - 7 pm
* Habitual napping (>20 minutes per day on a regular basis)
* Obliged to wake and care for family/friends (e.g. new born child etc)
* Use of antidepressants
* Depressed mood (Center of Epidemiologic Studies of Depression 20-item scale questionnaire)
* Travel arrangements outside time zone within the periods of data collection
* Travel arrangements outside time zone within period of intervention/control condition
* Inability to adhere to a sleep hygiene intervention/sleep schedule due to time commitments

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Sleep Duration | baseline
  Wrist Actigraphy
Sleep Duration | week 4
  Wrist Actigraphy
Sleep Quality | baseline
  Wrist Actigraphy
Sleep Quality | week 4
  Wrist Actigraphy

SECONDARY OUTCOMES:
BMI | baseline
BMI | day 28
Body fat percentage | baseline
Body fat percentage | day 28
Blood pressure | baseline
Blood pressure | day 28
Fasting blood glucose | baseline
Fasting blood glucose | day 28
Fasting total cholesterol | baseline
Fasting HDL cholesterol | baseline
Fasting LDL cholesterol | baseline
Fasting triglycerides | baseline
Fasting total cholesterol | day 28
Fasting HDL cholesterol | day 28
Fasting LDL cholesterol | day 28
Fasting triglycerides | day 28
plasma leptin | baseline
plasma leptin | day 28
plasma ghrelin | baseline
plasma ghrelin | day 28
plasma insulin | baseline
plasma insulin | day 28
plasma cortisol | baseline
plasma cortisol | day 28
Homeostasis model assessment estimated insulin resistance (HOMA-IR) | baseline
Homeostasis model assessment estimated insulin resistance (HOMA-IR) | day 28
Waist circumference | baseline
Waist circumference | day 28
Hip circumference | baseline
Hip circumference | day 28
Lean body mass | baseline
Lean body mass | day 28
Digital volume pulse - Stiffness Index (SI) | baseline
Digital volume pulse - Stiffness Index (SI) | day 28
Digital volume pulse - Reflection Index (RI) | baseline
Digital volume pulse - Reflection Index (RI) | day 28
Mnemonic Similarity Test (MST) | baseline
Mnemonic Similarity Test (MST) | day 28
Dietary Intake (7-day food diary) | baseline
Dietary Intake (7-day food diary) | week 4
Resting Metabolic Rate (RMR) | baseline
Resting Metabolic Rate (RMR) | day 28
Total Energy Expenditure (TEE) | baseline
Total Energy Expenditure (TEE) | day 21-23
Urinary 6-sulphatoxymelatonin | baseline
  Analysed from spot urine sample
Urinary 6-sulphatoxymelatonin | day 28
  Analysed from spot urine sample
Recent Physical Activity Questionnaire (RPAQ) | baseline
Recent Physical Activity Questionnaire (RPAQ) | day 28
Sleep Hygiene Index (SHI) | baseline
Sleep Hygiene Index (SHI) | day 28
Eating Choices Index (ECI) | baseline
Eating Choices Index (ECI) | day 28
Pittsburgh Sleep Quality Index (PSQI) | baseline
Pittsburgh Sleep Quality Index (PSQI) | day 28

OTHER OUTCOMES:
Dutch Eating Behaviour Questionnaire (DEBQ) | baseline
Women's Health Questionnaire | baseline
  Questionnaire to identify menstrual phase
Women's Health Questionnaire | day 21
  Questionnaire to identify menstrual phase

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Hall, PhD, Principal Investigator — King's College London
Locations (1):
- Diabetes & Nutritional Sciences Division, King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bosy-Westphal A, Hinrichs S, Jauch-Chara K, Hitze B, Later W, Wilms B, Settler U, Peters A, Kiosz D, Muller MJ. Influence of partial sleep deprivation on energy balance and insulin sensitivity in healthy women. Obes Facts. 2008;1(5):266-73. doi: 10.1159/000158874. Epub 2008 Oct 23. PMID 20054188
- [Background] Brondel L, Romer MA, Nougues PM, Touyarou P, Davenne D. Acute partial sleep deprivation increases food intake in healthy men. Am J Clin Nutr. 2010 Jun;91(6):1550-9. doi: 10.3945/ajcn.2009.28523. Epub 2010 Mar 31. PMID 20357041
- [Background] Buxton OM, Pavlova M, Reid EW, Wang W, Simonson DC, Adler GK. Sleep restriction for 1 week reduces insulin sensitivity in healthy men. Diabetes. 2010 Sep;59(9):2126-33. doi: 10.2337/db09-0699. Epub 2010 Jun 28. PMID 20585000
- [Background] Markwald RR, Melanson EL, Smith MR, Higgins J, Perreault L, Eckel RH, Wright KP Jr. Impact of insufficient sleep on total daily energy expenditure, food intake, and weight gain. Proc Natl Acad Sci U S A. 2013 Apr 2;110(14):5695-700. doi: 10.1073/pnas.1216951110. Epub 2013 Mar 11. PMID 23479616
- [Background] Shechter A, Rising R, Albu JB, St-Onge MP. Experimental sleep curtailment causes wake-dependent increases in 24-h energy expenditure as measured by whole-room indirect calorimetry. Am J Clin Nutr. 2013 Dec;98(6):1433-9. doi: 10.3945/ajcn.113.069427. Epub 2013 Oct 2. PMID 24088722
- [Background] Spiegel K, Leproult R, Van Cauter E. Impact of sleep debt on metabolic and endocrine function. Lancet. 1999 Oct 23;354(9188):1435-9. doi: 10.1016/S0140-6736(99)01376-8. PMID 10543671
- [Background] St-Onge MP, Roberts AL, Chen J, Kelleman M, O'Keeffe M, RoyChoudhury A, Jones PJ. Short sleep duration increases energy intakes but does not change energy expenditure in normal-weight individuals. Am J Clin Nutr. 2011 Aug;94(2):410-6. doi: 10.3945/ajcn.111.013904. Epub 2011 Jun 29. PMID 21715510
- [Background] St-Onge MP, O'Keeffe M, Roberts AL, RoyChoudhury A, Laferrere B. Short sleep duration, glucose dysregulation and hormonal regulation of appetite in men and women. Sleep. 2012 Nov 1;35(11):1503-10. doi: 10.5665/sleep.2198. PMID 23115399
- [Derived] Al Khatib HK, Hall WL, Creedon A, Ooi E, Masri T, McGowan L, Harding SV, Darzi J, Pot GK. Sleep extension is a feasible lifestyle intervention in free-living adults who are habitually short sleepers: a potential strategy for decreasing intake of free sugars? A randomized controlled pilot study. Am J Clin Nutr. 2018 Jan 1;107(1):43-53. doi: 10.1093/ajcn/nqx030. PMID 29381788
- See also: Primary publication — http://www.ncbi.nlm.nih.gov/pubmed/29381788